CLINICAL TRIAL: NCT01601145
Title: Effect of Probiotic on the Plaque pH. A Randomized Double Blind Interventional Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Università degli Studi di Sassari (Other)
Responsible Party: Principal Investigator, Guglielmo Campus, Associate Professor of Community Dentistry, Università degli Studi di Sassari
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 146/2011
Record Dates: First submitted 2012-05-15; First posted 2012-05-17 (Estimated); Last update posted 2012-08-22 (Estimated); Status verified 2012-08

CONDITIONS: Plaque Ph Lowering After Use of Probiotics; Caries; Gingivitis
Keywords: Lactobacillus Brevis CD2; schoolchildren; dental caries; Gingivatis
MeSH Terms: conditions — Gingivitis; Dental Caries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- lozenges with Lactobacillus brevis CD2 (Experimental): Randomized group using lozenges for 6 weeks.
  Interventions: Dietary Supplement: consumption of lozenges
- lozenges (Placebo Comparator): Randomized group using lozenges for 6 weeks.
  Interventions: Dietary Supplement: consumption of lozenges

INTERVENTIONS:
Dietary Supplement: consumption of lozenges — Each subject two lozenges a day for 6 weeks

SUMMARY:
The aim of the present research protocol was to evaluate the effect of probiotics daily used, on the plaque acidogenicity of children. The null hypothesis was that the plaque acidogenicity would remain unchanged and not associate with the use of probiotics. Moreover, the in situ study will be carried out to investigate the plaque formation as biofilm in demineralised enamel specimens following the regular consumption of a probiotic product compared to a control group. Metabolic of the biofilm formed on of the enamel specimens resulting from the consumption will be evaluated over a period of 8 weeks.

DETAILED DESCRIPTION:
Prior to the start of the study, demographic, ethnic and prognostic data will be collected (screening phase). A medical history will be taken, with documentation of previous and concomitant treatment and a clinical examination of the oral cavity (dental status, oral mucosa) will be performed by the investigator. If the test subject meets all the inclusion criteria without fulfilling any of the exclusion criteria, he/she will be enrolled in the clinical trial and given a test subject identification number.

All test subjects will receive a patient diary in the screening phase.

Washout phase I (1 week):

The test subjects will use only the fluoride-containing toothpaste provided by the sponsor for daily oral hygiene. A soft toothbrush will likewise be provided.

The test subjects will also receive a patient diary which will inform them that during the treatment phase they may not use any fluoride containing oral hygiene products (tooth-paste, mouthwashes, gels etc.) other than the study tooth-paste, drink any fluoride-containing mineral water or black tea, or eat any fish meals.

Treatment phase I (6 weeks):

Following washout phase I, the test subjects start the first treatment phase. Plaque pH measurements at 1 week.

All subjects are instructed about oral hygiene and about the consumption of the study product.

Treatment phase II (1 week after):

The test subjects will use only the fluoride-containing toothpaste provided by the sponsor for daily oral hygiene. A soft toothbrush will likewise be provided. Plaque pH measurements.

1. MATERIALS AND METHODS 1.1 Clinical parameters DMFT index, gingival index

   1.2 Investigation of saliva factors Saliva factors pH and flow rate will be measured during the screening phase on three days, each time in the morning. The mean of the three measurements will be calculated.

   The Dentobuff® test kit (Vivadent, Liechtenstein) will be used.

   1.3 Teeth brushing technique Test subjects are required to clean their teeth three times a day with the fluoride-containing toothpaste and a soft toothbrush. During that time, a fresh, damp gauze (soaked in water) will be placed in the container each day in order to provide a moist atmosphere for the appliances. The specimens should not be allowed to dry out.

   The enamel specimens themselves are likewise carefully cleaned with the soft toothbrush except the last day of every period.

   1.4 Randomization Using a computer program (Excel 2003 for Mac OsX), the randomization will carried out on an individual basis.

   1.5 Application of the study product The subjects are not allowed to chew the lozenges. They are allowed to swallow the lozenges.

   1.6 Plaque-pH evaluation At the end of each phase plaque acidogenicity will be assessed using the MicroTouch technique after a previous sucrose challenge. Evaluations of pH will be carried out at on each specimen. The pH will be measured in quintuplicate at 6 different time points: at baseline (before sucrose rinse) and 2, 5, 10, 20 and 30 min after a 1-min rinse with 10 ml 10% sucrose, using active movements.

   An iridium touch microelectrode (diameter 0.1 mm; Beetrode® NMPH-1, World Precision Instruments, Sarasota, Fla., USA, with a porous glass reference electrode (MERE 1, World Precision Instruments) will be used. A salt bridge will be created in a KCl (3 M) solution between the reference electrode and a finger of the subject. Before each session of pH evaluation, the electrode will be calibrated using buffer solution at pH 7.00 and 4.00.
2. STATISTICAL METHODS AND DETERMINATION OF SAMPLE SIZE 2.1 Planned Analysis Descriptive summary statistics will be computed for all parameters documented in the case report form (CRF).

Quantitative parameters will be described by seven-point scales with mean, standard deviation, median, quartiles, minimum and maximum. Absolute and relative frequencies will be given for qualitative variables. All descriptions will be done separately for treatment groups and visits.

The full statistical analysis including details such as methods of dealing with outliers, missing values, data under prohibited concomitant medication, prohibited nutrition or other possible irregularities will be fixed in a more detailed statistical analysis plan, which will be updated during a blind review of the data before applying the randomisation code to the data for the final analysis.

In order to ensure that the database accurately reflects the data reported in the CRF, a double data entry procedure (data entered by different staff in two separate data files) will be used. In addition to an electronic comparison of these two data files a validation of the data will check ranges, consistency and plausibility. Unclear data will undergo a data cleaning process ("queries"). Any changes applied to data in the database during data cleaning will be recorded in a special log file. The database will be frozen on completion of data cleaning.

Appropriate validated software (e.g. SAS, SPSS) will be used for the data processing and statistical evaluation.

Confirmative statistical testing For confirmative statistical testing an analysis of variance (ANOVA) model will be used as a global test, including the treatment sequences as "between subject factors" and the treatment conditions as "within subject factors".

The full analysis will be described in detail in a specific statistical analysis plan before unblinding the data.

Adjustment of type I error due to multiple testing is not necessary due to a prior ordering of the hypotheses. Hypothesis testing has to be stopped if a null-hypothesis may not be rejected at the 5% error level α. This procedure maintains a constant global level of α = 5%.

ELIGIBILITY:
Inclusion Criteria:

* Written declaration of informed consent signed by parents/guardian
* At least 20 teeth
* Good general health, as assessed by investigator
* Average oral hygiene (cleaning the teeth at least twice a day)
* Agreement of test subject not to use any oral hygiene products other than the test products and toothpaste provided for the duration of the study; the use of non-fluoridated oral hygiene agents is allowed.
* Flow rate of stimulated saliva ≥ 0.7 ml/min
* At least on caries active lesion (d/D>0)

Exclusion Criteria:

* Ongoing oral or dental treatment except for emergency treatment.
* Known allergic reaction to an oral hygiene product and/or medication and/or dental material previously used in the mouth or pharynx.
* Existing allergy to one of the components of the test products or the standard toothpaste.
* Pathological changes of the oral mucosa, e.g. acute ulcerating gingivitis, acute herpetic gingivostomatitis, recurrent aphthous ulceration or systemic illnesses with oral manifestations.
* Use of fluoride-containing products (pastes, mouthrinses) within the 14 days prior to the introduction of the intra-oral appliances.
* Use of fluoride-containing products: gels, tablets, varnishes, fillings etc. or of erosive broncholytics or antiasthmatics within 30 days prior to the introduction of the intra-oral specimen holder.
* Antibiotic therapy within the past six months.
* Any non-permitted therapy.

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 192 (Actual)
Dates: Start 2012-01; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Lower plaque acidogenicity | 2 months
  The regular consumption of probiotic will lead to a significantly lower plaque acidogenicity compared to a placebo. Regular oral hygiene is permitted.

CONTACTS AND LOCATIONS:
Overall Officials: Guglielmo Campus, Principal Investigator — University of Sassari, Dept of Surgery, Microsurgery and Medicine Sciences
Locations (1):
- University of Sassari, Dept of Surgery, Microsurtgery and Medicine Sciences, Sassari, SS, Italy

REFERENCES:
- [Derived] Campus G, Cocco F, Carta G, Cagetti MG, Simark-Mattson C, Strohmenger L, Lingstrom P. Effect of a daily dose of Lactobacillus brevis CD2 lozenges in high caries risk schoolchildren. Clin Oral Investig. 2014;18(2):555-61. doi: 10.1007/s00784-013-0980-9. Epub 2013 May 5. PMID 23644602